CLINICAL TRIAL: NCT02914652
Title: The Cardiopulmonary Effect of Inhaled Beta-2-agonists on Adult Ventrucular Septal Defect Patients With Persistant or Surgically Corrected Conditions - The VENTI Trial
Brief Title: The Cardiopulmonary Effect of Inhaled Beta-2-agonists on Adult Patients Born With Ventricular Septum Defects.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CERCA5
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2017-10

CONDITIONS: Ventricular Septal Defect
Keywords: Congenital Heart Disease; Ventricular Septal Defect; Beta-2-agonists; Surgery; Follow-up
MeSH Terms: conditions — Heart Septal Defects, Ventricular; Heart Defects, Congenital | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Operated VSD's (Experimental): Through the use of Electronic Patient Journal (EPJ), the investigators have identified a total of 182 children who underwent surgical closure of a congenital VSD at Aarhus University Hospital, Denmark between 1990 and 1995. After thorough review of all charts, 117 patients were excluded from participation. Exclusion criteria were coexistence of other congenital heart defects (n=89), associated syndromes, e.g. Down's (n=14), operation through a ventricular approach (n=7), missing chart (n=6) and documented arrhythmia requiring pacemaker (n=1). The remaining 68 patients represent a homogeneous group comparing surgeons, anaesthetists, surgical procedure and post-surgical period. A fraction of this group will be randomly selected for this trial, and receives salbutamol or norflouran, blinded.
  Interventions: Drug: Salbutamol; Drug: Norflouran (Placebo Evohaler(R) )
- Un-operated VSD's (Experimental): Using EPJ, this project identified a total of 481 children born between 1985 and 1998 who had a small VSD, confirmed through diagnosis codes, that was not closed, neither spontaneously nor surgically. Exclusion criteria were lack of medical record, suffering from coronary disease, other congenital cardiac abnormalities than VSD, spontaneous closure of the ventricular septal defect at inclusion date, magnetic implants, pregnancy, lack of Danish language skills, suffering from lung disease requiring continuous medical treatment. The remaining patients represent a homogenous group of patients with isolated persistent ventricular septal defects. A fraction of this group will be randomly selected for this trial, and receives salbutamol or norflouran, blinded.
  Interventions: Drug: Salbutamol; Drug: Norflouran (Placebo Evohaler(R) )
- Healthy controls (Experimental): Will function as a control group. Controls will be recruited through www.forsoegsperson.dk and www.sundhed.dk. Current group receives salbutamol or norflouran, blinded.
  Interventions: Drug: Salbutamol; Drug: Norflouran (Placebo Evohaler(R) )

INTERVENTIONS:
Drug: Salbutamol — Ventoline(R), inhalation spray, 0,1 mg/dose, 9 doses administered as coherent single doses.
  Other Names: Ventoline
Drug: Norflouran (Placebo Evohaler(R) ) — Placebo Evohaler(R) MDI, inhalation spray, 60 mg/dose, 9 doses administered as coherent single doses.
  Other Names: Placebo

SUMMARY:
The overall objective for this study is to test whether β2-agonists will affect the cardiopulmonary capacity of VSD-operated patients compared with un-operated VSD-patients and healthy age- and gender-matched controls.

DETAILED DESCRIPTION:
1. Background information

   1.1. Investigational product Ventoline® 0,1 mg/dosis inhalation spray.

   The active substance is Salbutamol. Salbutamol is a selective β2-agonist which induces relaxation of the bronchial smooth muscles. Common side effects experienced in 1-10% of chronic Ventoline® users are tachycardia, cephalgia and tremors. For more information about the product go to 12. Appendix 1 - Product summary, which holds the Danish product resume from The Danish Health and Medicines Authority.

   1.2 Background Grown-ups with congenital heart disease represent a constantly growing cohort (1,2), and with a birth prevalence of 2.62 per 1000 live birth, isolated ventricular septal defect (VSD) is the most frequent congenital cardiac malformation (3,4). For these patients short- and long-term follow-up studies have displayed low complication rates (5-7), and VSD-corrected patients have been assumed to be just as healthy and physically fit compared as their peers (8). Nevertheless recent studies have demonstrated significant long-term abnormalities (9-12).

   Compared with the normal population similar workloads in ergometer cycle test have been demonstrated in some studies (13-17) whereas other studies have observed subnormal working capacity in these VSD patients (18-20). The most recent study, demonstrated significantly lower cardiopulmonary exercise capacity (9), a lower force frequency response (10), and abnormal ventilation pattern compared with healthy age and gender matched controls (11). How the abnormal pulmonary function interrelates with the impaired cardiac function and the limited exercise capacity remains to be clarified. None of the referred studies have explained the mechanism for the impaired exercise capacity. However, chronotropic incompetence (9,14,15,19,21) due to postsynaptic β-adrenergic desensitization of the cardiac autonomic nervous system after corrective cardiac surgery (14,15,19,21) have been suggested. Intrinsic sinus node dysfunction in postoperative congenital heart disease patients has also been demonstrated and may explains the lower exercise capacity (22,23). Moreover, abnormal pulmonary function has been demonstrated in these patients, which may be due to a direct mechanical limitation to breathing caused by the sternotomy the patient underwent earlier in life. However, there may also be an indirect physiological explanation to the abnormal exercise ventilation. A previous study found that the pulmonary function was somewhat decreased in many of the standard parameters, perhaps pointing in the direction of a direct mechanical restriction, but without any clear results(24). The study lacks a reference group of healthy controls, using standardized pulmonary values instead. Moreover, the patient group only consisted of children, not adults, making it difficult to predict the long-term outcome in this group of patients.

   β-adrenoceptors in heart (β1) and lungs (β2) are targets for catecholamine's causing stimulation of the sympathetic nervous system with among other effects bronchodilation and positive chronotropic, dromotropic, and ionotropic effects in the heart (25). Inhaled β2-agonists are commonly used as bronchodilators for patients conditioned with increased airway resistance (26). It has long been discussed if they have an ergogenic potential in sport due to both the effects on the lungs and a theoretical effect on the heart. It is now well described that exercise performance and maximal oxygen uptake (VO2-max) are not affected in healthy adults (27-29) not even when supratherapeutic doses of salbutamol are tested (27). However, these studies were mainly performed in athletes and not on the general population. In patients with chronic cor pulmonale a moderate chronotropic effect from β2-agonist infusions have been demonstrated (30). The effect in patients with congenital heart disease such as VSD is unknown. Since the VSD patients have an impaired pulmonary function as well as an impact on their chronotropic and ionotropic function, they might benefit from treatment of β2-agonists.
2. Hypotheses

   A) Patients with surgically corrected VSD have an increased airway resistance at rest which is positively affected by inhaled β2-agonists.

   B) Patients with surgically corrected VSD have impaired spirometry outcomes which is positively affected by inhaled β2-agonists.

   C) Patients with surgically corrected VSD have an inferior diffusion lung capacity compared with un-operated VSD-patients and healthy controls.

   D) β2-agonists increase peak exercise minute ventilation and thereby the cardiopulmonary exercise capacity of surgically corrected VSD patients compared to un-operated VSD-patients and healthy controls.

   E) Inhaled β2-agonists increase peak exercise heart rate and thereby the cardiopulmonary exercise capacity of patients with surgically corrected VSD compared to un-operated VSD-patients and healthy controls.

   F) Patients with surgically corrected VSD have a reduced heart rate variability, compared with un-operated VSD-patients and healthy controls, that is positively affected by β2-agonists.
3. Trial design

   The intended study will be conducted as a randomized controlled blinded cross over study, on the two VSD groups, matched with an equivalent number of controls. When written informed consent is obtained from participants they will be included in the trial. They will undergo two test days with an interval of at least of 48 hours and maximal 14 days, to ensure complete physical recovery and comparable physical condition at the two tests.

   It will be randomized whether the participant receives the Ventoline or the placebo at their first or second test day. To ensure similar test performances, both the participants and monitoring staff will be blinded in regards to what they are testing. For further information regarding study population see Chapter "Study Design" and "Arms and Investigations".
4. Methods

   The tests below are described in the order that they are supposed to be conducted. Each test will be performed on both test days at Aarhus University Hospital, Skejby at The Department of Cardiothoracic and Vascular Surgery.

   4.1 Bioelectrical impedance analysis (Bioimpedance)

   The data collected are Total Body Water (TBW), Extracellular Fluid (ECF), Intracellular Fluid (ICF), Fat Free Mass (FFM) and Fat Mass (FM).

   4.2 Lung Clearance Index

   The equipment will analyse LCI 2,5 (LCI is defined as the cumulative expired volume (CEV) divided by the functional residual capacity (FRC) ), Scond (ventilation heterogeneity generated in the conductive lung zone) and Sacin (ventilation heterogeneity generated peripheral to the acinar entrance.

   4.3 Plethysmography (Static lung function)

   The equipment determine different lung parameters of which we will measure total lung capacity (TLC, liters), residual volume (RV, liters), functional residual capacity (FRCpleth, ml) and specific airway resistance (sRAW, kPa/sec) (35).

   4.4 Spirometry

   The test will include forced expiratory volume in one second (FEV1), forced vital capacity (FVC), the ratio between the two volumes (FEV1/FVC) and peak expiratory flow (PEF).

   4.5 Diffusion capacity test

   The diffusion capacity test will be performed on the same equipment as the plethysmography. The test determines lung carbon monoxide diffusion capacity (DLCO) and alveolar volume (VA) expressed as percentage of expected value.

   4.6 Impulse oscillometry

   The equipment will then be able to analyse resistance in of the respiratory system at 5 Hz (R5), and at 20 Hz (R20) and the difference between the two measured resistances (Diff 5-20) (38,39).

   4.7 Holter-Monitorisation

   ECG activity during and after orthostatic and exercise testing will be monitored with a 2-channel Holter monitor. Participants will be wearing the Holter-Monitors for 48 hours after activation at the first visit and for 24 hours after activation at the second visit. This results in 3 data-files:

   With the Pathfinder analysis software, we will assess any ECG changes and heart rate variability (HRV) during and after each exercise test. Endpoints are HRV (beat-to-beat variation) and mediterranean hour pulse.

   4.8 Orthostatic stress test (active standing)

   During the test we will measure blood pressure and heart rate with an automated sphygmomanometer on the left forearm.

   4.9 Exercise testing

   Exercise capacity will be tested on a Lode Corival ® ergometer cycle. With the Jaeger MaesterScreen CPX software system, we will monitor pulmonary ventilation and gas exchange in a breath-by-breath measurement. During test sessions, heart rate, blood pressure and electrocardiogram, will be measured continuously. The Holter-monitor is also recording during the exercise test.

   Each test day lasts approximately 4-5 hours.
5. Statistics

   If suitable, continuous data will be reported as mean ± standard deviation (SD), otherwise they will be displayed as median value with 95% confidence intervals (CIs). Comparison of continuous data will be by unpaired Student's t-tests or, for non-normal-distributed data, the Mann-Whitney-Wilcoxon rank sum test. All correlations will be checked with simple regression analyses. Data from all included participants will be used for the statistical analyse. If correlations are made with the data material it will be evident on the published material. Data analysis will be performed with Stata/ IC 12.1 for Mac (StataCorp, Texas, United States of America).

   5.1. Power calculation

   Our main hypothesis is that β2-agonists increase peak exercise oxygen uptake to the same level as healthy controls. Previously, the same cohort of VSD patients was exercise tested in another study and in terms of peak oxygen uptake a statistically and clinically significant difference was found compared with controls; 38.0 ± 8.2 ml kg-1 min-1 vs. 47.7 ± 6.5 ml kg-1 min-1 9. If we assume a true difference of approximately 75% with the current endpoint, and apply a statistical power of 90 % and a level of significance of 95 %, we therefore need to include 26 participants in each of the three group. We aim at including 30 participants in each group and a total study population of 90 participants.

   Deviations in the statistics or power calculation will be evident in in published material.
6. Data storage

   Each participant will be given an identification number used for all purposes. A list over identification codes and complete name, address and telephone number will be saved and securely stored with the Trial Master File (TMF) and in REDCap. Data will be stored for 10 years. All digitalised data will be stored on two harddrives - one portable external harddrive that is kept safe behind two locked doors at the department and one external server named REDCap with continous back-up. Each identification number will have a Case Report Form (CRF) that also holds printed trial documents. Physical documents will be stored behind two locked doors and the CRF will be stored with the TMF.

   A source datasheet for the information noted in the CRF will be stored with the TMF. It will hold information on the origin of source data concerning, inclusion and exclusion, randomisation, bioimpedance data, Lung function data, Holter-Recordings and Holter-Recording analyses data, orthostatic stress test data and Exercise testing data.
7. Ethical concerns

The study is conducted in accordance with the Helsinki declaration and Danish law.

The project will obtain permission from the Danish Protection Agency, the Danish Health and Medicines Authority, and The Central Denmark Region Committees on Health Research Ethics. Data will be handled in agreement with the personal data handling law and the participants' safety is always the number one priority during this trial.

The project will be supervised by the department of Good Clinical Practice (the GCP-Unit).

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age and legally competent to vouch for their own study participation.
* Informed and written consent for participation in this trial.
* Trial group 1: Surgically corrected for isolated VSD between 1990 and 1998 at Aarhus University Hospital.
* Trial group 2: Diagnosed with isolated VSD born between 1985 and 1998 without surgical or percutaneous closure. Verified by Echocardiography within the last 4 years. If it is more than 4 it will be verified by our doctors as a systolic murmur or echocardiography.
* Trial group 3: 18-30 years, with no known medical records of heart and lung disease.
* Restrain from strenuous leg exercise 24 hours before inclusion.

Exclusion Criteria:

* Lack of medical record.
* Pregnancy.

  o Participants will be asked if they are using contraceptives and be told to continue this during the trial and for at least 30 hours (5 times T2) after their last visit. If they are not using spiral or valid contraceptives (contraceptive pills, implants, transdermal patches, vaginal ring or injections) one of our medical experts will judge if the participant is able to undergo the trial. They will likewise be informed to withstand from sexual intercourse during the trial until 30 hours after the second visit.
* Currently breastfeeding.
* Syndromes, such as Down's.
* Mentally or physically incompetent to perform the ergometer bicycle test.
* Thyrotoxicosis.
* Pre-trial medical record of arrhythmias except right bundle branch block.
* Asthma or other known β2-responsive conditions.
* Coronary heart disease.
* Severe pulmonary disease.
* Diabetes.
* Use of the following medication: Xantin-derivates, steroids, diuretics, ipratropium.
* Allergy to the active ingredients of Ventoline: Salbutamolsulphate, benzalkoniumchloride

The product summary was used to establish exclusion criteria in regards to medication and diseases that aren't eligible with the medical treatment. Other medication than described in the in- and exclusion criteria will be noted in the participants CRF. If the participant takes any special medication one of our trial doctors will determine if the participant should be excluded.

Participants will be informed of the exclusion criteria in the information letter and at the initial information interview before inclusion in the trial. Oral verification is considered sufficient to verify the exclusion criteria.

Ages: 21 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Minute Ventilation (ml/min) in VSD-operated patientes | 21 to 26 years after surgical closure.
Peek Exercise Oxygen Uptake (ml O2/kg/min) in VSD-operated patientes | 21 to 26 years after surgical closure.
Maximal workload (W) in VSD-operated patientes. | 21 to 26 years after surgical closure.

SECONDARY OUTCOMES:
Peak heart rate at maximal exercise, in VSD-operated patients. | Twentyone to 26 years after surgical closure.
Forced expiratory volume in 1 second (FEV1), in VSD-operated patients. | 21 to 26 years after surgical closure.
Airway resistance (R5-R20), in VSD-operated patients. | 21 to 26 years after surgical closure.
Hear-rate variability, in VSD-operated patients. | 21 to 26 years after surgical closure.
Diffusion capacity (DLCO), in VSD-operated patients. | 21 to 26 years after surgical closure.
Alveolar volume, in VSD-operated patients. | 21 to 26 years after surgical closure.
Lung clearance index, in VSD-operated patients. | 21 to 26 years after surgical closure.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, MD PhD DMSc, Principal Investigator — Dept. of Cardiothoracic & Vascular Surgery, Aarhus University Hospital, Skejby
Locations (1):
- Dept. of Cardiothoracic and Vascular Surgery, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Dolk H, Loane M, Garne E; European Surveillance of Congenital Anomalies (EUROCAT) Working Group. Congenital heart defects in Europe: prevalence and perinatal mortality, 2000 to 2005. Circulation. 2011 Mar 1;123(8):841-9. doi: 10.1161/CIRCULATIONAHA.110.958405. Epub 2011 Feb 14. PMID 21321151
- [Background] Warnes CA, Liberthson R, Danielson GK, Dore A, Harris L, Hoffman JI, Somerville J, Williams RG, Webb GD. Task force 1: the changing profile of congenital heart disease in adult life. J Am Coll Cardiol. 2001 Apr;37(5):1170-5. doi: 10.1016/s0735-1097(01)01272-4. No abstract available. PMID 11300418
- [Background] van der Linde D, Konings EE, Slager MA, Witsenburg M, Helbing WA, Takkenberg JJ, Roos-Hesselink JW. Birth prevalence of congenital heart disease worldwide: a systematic review and meta-analysis. J Am Coll Cardiol. 2011 Nov 15;58(21):2241-7. doi: 10.1016/j.jacc.2011.08.025. PMID 22078432
- [Background] Marelli AJ, Mackie AS, Ionescu-Ittu R, Rahme E, Pilote L. Congenital heart disease in the general population: changing prevalence and age distribution. Circulation. 2007 Jan 16;115(2):163-72. doi: 10.1161/CIRCULATIONAHA.106.627224. Epub 2007 Jan 8. PMID 17210844
- [Background] Penny DJ, Vick GW 3rd. Ventricular septal defect. Lancet. 2011 Mar 26;377(9771):1103-12. doi: 10.1016/S0140-6736(10)61339-6. Epub 2011 Feb 23. PMID 21349577
- [Background] Bol-Raap G, Weerheim J, Kappetein AP, Witsenburg M, Bogers AJ. Follow-up after surgical closure of congenital ventricular septal defect. Eur J Cardiothorac Surg. 2003 Oct;24(4):511-5. doi: 10.1016/s1010-7940(03)00430-5. PMID 14500067
- [Background] Roos-Hesselink JW, Meijboom FJ, Spitaels SE, Van Domburg R, Van Rijen EH, Utens EM, Bogers AJ, Simoons ML. Outcome of patients after surgical closure of ventricular septal defect at young age: longitudinal follow-up of 22-34 years. Eur Heart J. 2004 Jun;25(12):1057-62. doi: 10.1016/j.ehj.2004.04.012. PMID 15191777
- [Background] Menting ME, Cuypers JA, Opic P, Utens EM, Witsenburg M, van den Bosch AE, van Domburg RT, Meijboom FJ, Boersma E, Bogers AJ, Roos-Hesselink JW. The unnatural history of the ventricular septal defect: outcome up to 40 years after surgical closure. J Am Coll Cardiol. 2015 May 12;65(18):1941-51. doi: 10.1016/j.jacc.2015.02.055. PMID 25953746
- [Background] Heiberg J, Laustsen S, Petersen AK, Hjortdal VE. Reduced long-term exercise capacity in young adults operated for ventricular septal defect. Cardiol Young. 2015 Feb;25(2):281-7. doi: 10.1017/S1047951113002084. Epub 2013 Nov 21. PMID 24565413
- [Background] Heiberg J, Schmidt MR, Redington A, Hjortdal VE. Disrupted right ventricular force-frequency relationships in adults operated for ventricular septal defect as toddlers: abnormal peak force predicts peak oxygen uptake during exercise. Int J Cardiol. 2014 Dec 20;177(3):918-24. doi: 10.1016/j.ijcard.2014.10.009. Epub 2014 Oct 28. PMID 25456699
- [Background] Heiberg J, Petersen AK, Laustsen S, Hjortdal VE. Abnormal ventilatory response to exercise in young adults operated for ventricular septal defect in early childhood: A long-term follow-up. Int J Cardiol. 2015 Sep 1;194:2-6. doi: 10.1016/j.ijcard.2015.05.071. Epub 2015 May 15. PMID 26011258
- [Background] Heiberg J, Ringgaard S, Schmidt MR, Redington A, Hjortdal VE. Structural and functional alterations of the right ventricle are common in adults operated for ventricular septal defect as toddlers. Eur Heart J Cardiovasc Imaging. 2015 May;16(5):483-9. doi: 10.1093/ehjci/jeu292. Epub 2014 Dec 31. PMID 25552465
- [Background] Meijboom F, Szatmari A, Utens E, Deckers JW, Roelandt JR, Bos E, Hess J. Long-term follow-up after surgical closure of ventricular septal defect in infancy and childhood. J Am Coll Cardiol. 1994 Nov 1;24(5):1358-64. doi: 10.1016/0735-1097(94)90120-1. PMID 7930261
- [Background] Norozi K, Gravenhorst V, Hobbiebrunken E, Wessel A. Normality of cardiopulmonary capacity in children operated on to correct congenital heart defects. Arch Pediatr Adolesc Med. 2005 Nov;159(11):1063-8. doi: 10.1001/archpedi.159.11.1063. PMID 16275798
- [Background] Binkhorst M, van de Belt T, de Hoog M, van Dijk A, Schokking M, Hopman M. Exercise capacity and participation of children with a ventricular septal defect. Am J Cardiol. 2008 Oct 15;102(8):1079-84. doi: 10.1016/j.amjcard.2008.05.063. Epub 2008 Jul 26. PMID 18929713
- [Background] Hovels-Gurich HH, Konrad K, Skorzenski D, Nacken C, Minkenberg R, Messmer BJ, Seghaye MC. Long-term neurodevelopmental outcome and exercise capacity after corrective surgery for tetralogy of Fallot or ventricular septal defect in infancy. Ann Thorac Surg. 2006 Mar;81(3):958-66. doi: 10.1016/j.athoracsur.2005.09.010. PMID 16488701
- [Background] Cumming GR. Maximal exercise capacity of children with heart defects. Am J Cardiol. 1981 Jun;47(6):1381. doi: 10.1016/0002-9149(81)90273-3. No abstract available. PMID 7234707
- [Background] Otterstad JE, Simonsen S, Erikssen J. Hemodynamic findings at rest and during mild supine exercise in adults with isolated, uncomplicated ventricular septal defects. Circulation. 1985 Apr;71(4):650-62. doi: 10.1161/01.cir.71.4.650. PMID 3971536
- [Background] Pieroni DR, Nishimura RA, Bierman FZ, Colan SD, Kaufman S, Sanders SP, Seward JB, Tajik AJ, Wiggins JW, Zahka KG. Second natural history study of congenital heart defects. Ventricular septal defect: echocardiography. Circulation. 1993 Feb;87(2 Suppl):I80-8. PMID 8425326
- [Background] Reybrouck T, Rogers R, Weymans M, Dumoulin M, Vanhove M, Daenen W, Van der Hauwaert L, Gewillig M. Serial cardiorespiratory exercise testing in patients with congenital heart disease. Eur J Pediatr. 1995 Oct;154(10):801-6. doi: 10.1007/BF01959785. PMID 8529676
- [Background] Perrault H, Drblik SP, Montigny M, Davignon A, Lamarre A, Chartrand C, Stanley P. Comparison of cardiovascular adjustments to exercise in adolescents 8 to 15 years of age after correction of tetralogy of fallot, ventricular septal defect or atrial septal defect. Am J Cardiol. 1989 Jul 15;64(3):213-7. doi: 10.1016/0002-9149(89)90460-8. PMID 2741830
- [Background] Norozi K, Wessel A, Alpers V, Arnhold JO, Binder L, Geyer S, Zoege M, Buchhorn R. Chronotropic incompetence in adolescents and adults with congenital heart disease after cardiac surgery. J Card Fail. 2007 May;13(4):263-8. doi: 10.1016/j.cardfail.2006.12.002. PMID 17517345
- [Background] Ohuchi H, Watanabe K, Kishiki K, Wakisaka Y, Echigo S. Heart rate dynamics during and after exercise in postoperative congenital heart disease patients. Their relation to cardiac autonomic nervous activity and intrinsic sinus node dysfunction. Am Heart J. 2007 Jul;154(1):165-71. doi: 10.1016/j.ahj.2007.03.031. PMID 17584572
- [Background] Sulc J, Samanek M, Zapletal A, Voriskova M, Hucin B, Skovranek J. Lung function in VSD patients after corrective heart surgery. Pediatr Cardiol. 1996 Jan-Feb;17(1):1-6. doi: 10.1007/BF02505804. PMID 8778695
- [Background] Baker JG. The selectivity of beta-adrenoceptor agonists at human beta1-, beta2- and beta3-adrenoceptors. Br J Pharmacol. 2010 Jul;160(5):1048-61. doi: 10.1111/j.1476-5381.2010.00754.x. PMID 20590599
- [Background] Lehmann S, Bakke PS, Eide GE, Gulsvik A. Bronchodilator response to adrenergic beta2-agonists: relationship to symptoms in an adult community. Respir Med. 2007 Jun;101(6):1183-90. doi: 10.1016/j.rmed.2006.11.007. Epub 2006 Dec 22. PMID 17188486
- [Background] Kindermann W. Do inhaled beta(2)-agonists have an ergogenic potential in non-asthmatic competitive athletes? Sports Med. 2007;37(2):95-102. doi: 10.2165/00007256-200737020-00001. PMID 17241101
- [Background] Pluim BM, de Hon O, Staal JB, Limpens J, Kuipers H, Overbeek SE, Zwinderman AH, Scholten RJ. beta(2)-Agonists and physical performance: a systematic review and meta-analysis of randomized controlled trials. Sports Med. 2011 Jan 1;41(1):39-57. doi: 10.2165/11537540-000000000-00000. PMID 21142283
- [Background] Morton AR, Joyce K, Papalia SM, Carroll NG, Fitch KD. Is salmeterol ergogenic? Clin J Sport Med. 1996 Oct;6(4):220-5. doi: 10.1097/00042752-199610000-00003. PMID 8894333
- [Background] Vik-Mo H, Halvorsen FJ, Thorsen E, Walde NH, Rosland GA. Improved cardiac performance by salbutamol, a selective beta 2-agonist, in chronic cor pulmonale. J Cardiovasc Pharmacol. 1987 Feb;9(2):129-34. doi: 10.1097/00005344-198702000-00001. PMID 2435988
- [Derived] Eckerstrom F, Rex CE, Maagaard M, Rubak S, Hjortdal VE, Heiberg J. Exercise performance after salbutamol inhalation in non-asthmatic, non-athlete individuals: a randomised, controlled, cross-over trial. BMJ Open Sport Exerc Med. 2018 Aug 30;4(1):e000397. doi: 10.1136/bmjsem-2018-000397. eCollection 2018. PMID 30233808